CLINICAL TRIAL: NCT04766372
Title: A Multi-component Physical Activity Intervention for Adolescent Girls: Feasibility Cluster Randomised Controlled Trial
Brief Title: A Multi-component Physical Activity Intervention for Adolescent Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Dublin City University (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HERizonProject2
Record Dates: First submitted 2021-02-15; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Exercise
Keywords: physical activity; adolescent girls; feasibility; behaviour change
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Using block randomisation on Microsoft Excel, participants will be assigned to one of the four groups following baseline measures
Masking Description: Due to the nature of the study, it will not be possible to blind participants to their study condition (as they will know whether they are engaging the physical activity programme or not). As the researchers will be doing the data collection and conducting the behaviour change support calls, it will also not be possible to blind the researcher to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Menu of physical activity options (Experimental): Participants in all 4 groups will receive this booklet with suggestions of ways to be physically active, e.g. YouTube workouts, cycling or jogging, sports, or design their own using a home-based exercise booklet. Participants are asked to do 3 exercise sessions of 30 minutes per week. Participants are asked to record what activity they did and the duration of the session using a method most convenient for them, e.g. notes on their phone, wall calendar or using an activity log template which we will provide.
  .
  Interventions: Other: Behaviour change
- Physical activity programme (Experimental): Participants in the second group with receive the activity menu (as described above) as well as a detailed physical activity programme. This programme includes supportive weekly text messages, access to live workouts and access to an online social community.
  Interventions: Other: Behaviour change
- Individual behaviour change support (Experimental): Participants in the third group with receive the activity menu (as described above) as well as individual behaviour change support. Each participant is partnered with a trainee sport psychology ("Activity Mentor") who they have weekly video calls with to support their health behaviour change.
  Interventions: Other: Behaviour change
- Activity Programme & Behaviour Change Support (Experimental): Participants in the fourth group will receive all of the above (exercise menu, live workouts, social community, support texts and weekly calls with an Activity Mentor).
  Interventions: Other: Behaviour change

INTERVENTIONS:
Other: Behaviour change — Using needs supportive, self-determination theory-based, components to improve the physical activity behaviours of adolescent girls.

SUMMARY:
A four-arm randomised pilot trial involving:

1. Physical activity programme only - live exercise sessions, social support, standardised text messages
2. Individual behaviour change support only - regular one-to-one video calls with an activity mentor
3. Combined - Physical activity provision and individual behaviour change support
4. Usual care control All groups will be provided with a menu of physical activities.

Objectives.

To conduct a RE-AIM evaluation of a 6-month multi-component PA intervention for adolescent girls, through investigating:

* Who the intervention reaches, how representative they are for the population (Reach, Adoption) and who is most likely to benefit from the intervention (Reach);
* The extent to which the intervention is delivered as intended (Implementation), and factors that affect this (Adoption);
* Preliminary impact on participants' PA, sedentary behaviour, cardiovascular fitness and psychological wellbeing at 3, 6 and 12 months (Effectiveness, Maintenance);
* The qualitatively examine the acceptability of the intervention for adolescent girls, and identify necessary refinements;
* To gather data to inform a sample size calculation for a main trail

DETAILED DESCRIPTION:
Procedures. Following written informed assent of participants and consent of parents/guardians, the researcher will have a short introductory video call with the participant and parent to talk through the next steps, give instructions on how to complete fitness tests and answer any questions. After this introduction, participants can carry out their fitness testing at home remotely under the supervision of the researcher (via Zoom) or their parent. Following written consent, participants will complete all questionnaires online (approximately 15 minutes) - self-reported physical activity, sociodemographic and psychosocial measures (behavioural regulation in exercise questionnaire, body-appreciation scale and self-esteem scale - details of each listed below). Participants will then complete the fitness measures using the Resistance Training for Teens (RTFT) app (30 minutes) - 20m shuttle run tests, long jump and push up test. Participants will wear an Actigraph accelerometer on their don-dominant wrist continuously, as outlined in the study protocol, for 9 days before starting their 12-week physical activity programme. In total, assessments should take approximately one hour and will be conducted at baseline (week 0), post-intervention (week 12) and follow up (week 24).

Randomisation. Participants will be randomly allocated to one of the four intervention arms following baseline measures. 40 participants will be allocated to each arm using block randomisation on Microsoft Excel.

Intervention group - The goals of this physical activity intervention are to 1) increase adolescent girls total physical activity levels and 2) improve adolescent girls health behaviours, including body appreciation and motivation. This study hopes to build on our prior feasibility work to help us to understand which components of the intervention are most effective, i.e. a physical activity programme, individual behaviour change support or a combination. To achieve these goals the following elements will be implemented:

* Menu of physical activity options: Participants in all four groups will be given a booklet with suggestions of ways to be physically active, e.g. YouTube workouts, cycling or jogging, sports, or design their own using a home-based exercise booklet. They are asked to do 3 sessions of 30 minutes per week. Participants are asked to record what activity they did and the duration of the session using a method most convenient for them, e.g. notes on their phone, wall calendar or using an activity log template which the investigators will provide.
* Physical activity programme: Participants in groups 1 and 3 will receive -

  * Non Reply SMS: Sent to the participant mobile three times per week by the primary researcher, Emma Cowley PhD candidate, from an online non-reply messaging service. This service is password protected. All messages will be standardised (not personally tailored) and will be focused on behaviour change techniques or reminders.
  * Live exercise sessions: The researcher (with personal training and physical education teaching qualifications) will host two online group fitness classes each week which participants are also invited to join. This option is to allow participants the potential to engage with the other participants on the programme from the comfort of their own homes. It is also thought that having a scheduled set time to join a class on line may increase motivation and improve adherence, however the choice to join the class is optional. From previous feasibility work, these sessions were a highlight of the programme and often times parents and siblings would join in too. Participants are invited to turn their cameras on for the intro and warm up, however this is not mandatory.
  * Access to a social media group: With participant and parental consent, participants are invited to join a private group community online where they can access additional resources provided by the research team, ask questions in an informal setting and communicate with the other participants in the programme. It is well researched that social connection is a facilitator to adolescent girls participation in physical activity and as participants will be exercising from home the investigators feel giving them access to a social, safe and virtual community can help give them this social connectedness to other adolescent girls of the same age. This is not compulsory and participants are free to join the group, leave the group or decline being added to the group without it affecting their participation in the rest of the programme.
* Individual behaviour change support:

  * Participants in group 2 and 3 will be partnered with an 'activity mentor' whom they will work with for the duration of the intervention. These activity mentors are postgraduate students either studying for an MSc in sport and exercise psychology, or post-MSc and undertaking professional training. Their role is to support the participants with improving their health behaviours, autonomy and motivation. Participants will receive weekly calls from week 0-6 and then calls on week 9 and 12. Calls will be via phone call, FaceTime or Teams video call. Behaviour change support will be based on self-determination theory principles (autonomy, competence and relatedness; Ryan & Deci, 2000). Each call will be based on a pre-planned session outline and will be goal orientated, participant centred and focused on physical activity. Calls are expected to last 10-20 minutes per participant. A sub-sample of calls will be audio recorded to assess intervention fidelity.

Control: menu of physical activity options only. As this project runs for 6 months it will not be possible to provide the control group with the full physical activity programme (this is part of a PhD study). However, it is intended to provide the control group participants with intervention materials (home-HIIT booklets, field-based testing instructions) so that participants can implement the physical activity programme without the direct oversight of the research team. At the end of the intervention, control participants will also be offered to do a group behaviour change psychology session with an activity mentor.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 13-16 years
* Living in the UK or Ireland
* Would like support with becoming more physically active
* Ability to participate in moderate intensity physical activity according to the Physical Activity Readiness Questionnaire

Exclusion Criteria:

* Have taken part in previous HERizon study
* Currently doing more than 1 hour of exercise or sport every day.
* Currently pregnant
* Not having access to at least ONE of the following: a smartphone, home computer, or parent smartphone.

Ages: 13 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in objective physical activity levels | Baseline to post-intervention (week 12)
  Participants objective PA will be monitored continuously (i.e. 24 h/day) over a nine-day period using an accelerometer (actigraph GT9x software). This device will be worn on their non-dominant wrist and uses the same validated MEMS sensor as the Actigraph GT3X+ model which has been validated (Hanggi et al., 2013) and used extensively with adolescents (Corder et al., 2016). Using the Actigraph, total daily PA, moderate-to-vigorous PA and sedentary time can be assessed.

SECONDARY OUTCOMES:
Aerobic capacity | week 0, week 12, week 24
  Measured by the 20m shuttle run test which has been validated as an effective instrument for adolescent aerobic capacity (Boreham et al., 1990). Participants will require 20m space e.g. garden or green space. Using the Resistance Training for Teens mobile app, participants will be given written and visual instructions of how to set up and perform the test. Participants are required to run back and forth between two markers (20m distance) on the sound of a beep. The audio can be played through the app.
Upper body strength | week 0, week 12, week 24
  Participants will do a push up test to the cadence of an audio recording. As above, written and visual instructions on how to set up and perform the test are provided on the app, as well as the audio file which sets the push up cadence. Should participants not be able to do a full push up (starting in high plank on hands and toes), they can lower onto their knees. It is important that the push up variation they choose is the same for baseline and post-intervention for fair comparison. No equipment is needed.
Strength/ Power | week 0, week 12, week 24
  Participants will do a long jump to assess their strength/power. They will start from one marker and just as far as they can and mark where they land. They will use a measuring tape to record this distance. If they do not have a measuring tape they can use their feet to measure and do this again for the post-intervention assessment for consistency. Again, the Resistance Training for Teens app provides visual and written instructions on set up and how to perform.
Change in Physical Activity Motivation | week 0, week 12, week 24
  measured by the 19-item Behavioural Regulation in Exercise Questionnaire (BREQ3) (Markland and Tobin, 2004) plus an additional five-items (Wilson et al., 2006). Using a 5 point Likert scale, the maximum score is 5 which indicates a high level of that particular sub-scale of motivation, e.g. intrinsic motivation rr amotivation.
Change in Body Appreciation | week 0, week 12, week 24
  measured by the 10-item Body Appreciation Scale (Avalos et al., 2005). Using a 5-point Likert scale, the maximum score is 5 which indicates a high level of body appreciation.
Change in Physical Activity Competence | week 0, week 12, week 24
  measured by the 4-item Perceived Competence Scale (Matsui & Muratas, 1997). Using a 7-point Likert scale, the maximum score is 7 which indicates a high level of competence towards physical activity.
Change in Self-esteeem | week 0, week 12, week 24
  measured by the 12-item Adolescent Self-Esteem Questionnaire (Hafekost et al., 2017). Using a 5-point Likert scale, the maximum score is 5 which indicates a high level of self-esteem
Change in objective physical activity levels | Baseline to follow-up (week 24)
  Participants objective PA will be monitored continuously (i.e. 24 h/day) over a nine-day period using an accelerometer (actigraph GT9x software). This device will be worn on their non-dominant wrist and uses the same validated MEMS sensor as the Actigraph GT3X+ model which has been validated (Hanggi et al., 2013) and used extensively with adolescents (Corder et al., 2016). Using the Actigraph, total daily PA, moderate-to-vigorous PA and sedentary time can be assessed.

OTHER OUTCOMES:
Process Evaluation | week 0, week 12, week 24
  Using a mixed methods approach, this study aims to conduct an evaluation of this physical activity intervention across five different domains (R-reach, E-effectiveness, A-adoption, I-implementation and M-maintenance).

CONTACTS AND LOCATIONS:
Overall Officials: Anton Wagenmakers, PhD, Principal Investigator — Liverpool John Moores University
Locations (3):
- Dublin City University, Dublin, Ireland
- United Kingdom (2):
  - Liverpool John Moores University, Liverpool, Merseyside
  - University of Liverpool, Liverpool

IPD SHARING:
Plan to Share IPD: No
We will use participant personal data in the ways needed to conduct and analyse the study and if necessary, to verify and defend, when required, the process and outcomes of the study. Personal data will be accessible to the study team. In addition, responsible members of Liverpool John Moores University be given access to personal data for monitoring and/or audit of the study to ensure that the study is complying with applicable regulations. When we do not need to use personal data, it will be deleted or identifiers will be removed. Consent form, contact details, audio recordings etc. will be retained for 10 years. We will not tell anyone that she has taken part in an interview. She will not be identifiable in any ensuing reports or publications.

REFERENCES:
- [Background] Cowley ES, Watson PM, Foweather L, Belton S, Thompson A, Thijssen D, Wagenmakers AJM. "Girls Aren't Meant to Exercise": Perceived Influences on Physical Activity among Adolescent Girls-The HERizon Project. Children (Basel). 2021 Jan 7;8(1):31. doi: 10.3390/children8010031. PMID 33430413
- [Background] Cowley ES, Watson PM, Foweather L, Belton S, Mansfield C, Whitcomb-Khan G, Cacciatore I, Thompson A, Thijssen D, Wagenmakers AJM. Formative Evaluation of a Home-Based Physical Activity Intervention for Adolescent Girls-The HERizon Project: A Randomised Controlled Trial. Children (Basel). 2021 Jan 22;8(2):76. doi: 10.3390/children8020076. PMID 33499174